CLINICAL TRIAL: NCT01053312
Title: A Principal, Open-Label, Single Center Study to Validate the Detection of Cerebral Cortical Amyloid With Flutemetamol (18F) Injection in Subjects Previously Biopsied
Brief Title: PET Imaging of Brain Amyloid in Normal Pressure Hydrocephalus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: i3 Statprobe (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GE 067-008
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Results first posted 2012-06-05 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: Amyloid; NPH Normal pressure hydrocephalus; PET Positron Emission Tomography; SUVR Standard uptake value ratios
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Alzheimer Disease | interventions — flutemetamol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 flutemetamol (Experimental)
  Interventions: Drug: [18F] Flutemetamol

INTERVENTIONS:
Drug: [18F] Flutemetamol — All subjects will receive an intravenous (IV) dose of [18F]flutemetamol (less than 10µg flutemetamol). The nominal activity of a single administration of [18F]flutemetamol will be 185 megabecquerels (MBq).
  Other Names: Flutemetamol; AH110690

SUMMARY:
This study will determine the level of association between the quantitative estimates of brain uptake of [18F]flutemetamol and the quantitative immunohistochemical estimates of amyloid levels in biopsy samples previously obtained during shunt placement in patients who have normal pressure hydrocephalus (NPH).

ELIGIBILITY:
Inclusion Criteria:

* The subject is 50 years old or older.
* The subject has had a frontal lobe cortical biopsy adequate for the detection and quantitation of amyloid.
* Informed consent has been signed and dated by the subject/and/or subjects' legally acceptable representative, if applicable, in accordance with local regulations.

Exclusion Criteria:

* The subject has a contraindication for MRI or PET.
* The subject has a known or suspected hypersensitivity/allergy to [18F]flutemetamol.
* The subject has participated in any clinical study using an investigational agent within 30 days of dosing.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-12; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim A Mansfield, MS, Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Flutemetamol Injection: [18F]flutemetamol (less than 10µg flutemetamol). The nominal activity of a single administration of [18F]flutemetamol will be 185 megabecquerels(MBq).
Period: Overall Study
Arm/Group | Flutemetamol Injection
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Flutemetamol Injection
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 70 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Estimates of Brain Uptake [18F]Flutemetamol and the Quantitative Immunohistochemical (IHC) Estimates of Amyloid Levels in Biopsy Samples Previously Obtained.
Description: Radiotracers have enabled the in-vivo imaging of amyloid-beta plaques in the brain, one of the histopathologic hallmarks of Alzheimer's disease (AD). Standardized uptake value ratio SUVR)is the quantitive measure of specific tracer uptake, normalized for the non-specific mean uptake in a reference region. SUVR is calculated as SUV_voi/SUV_ref with SUV being the integrated activity over a given time period for the volume of interest (SUV_voi) or reference region (SUV_ref). VOI means volume of interest and REF means reference region.
Time Frame: Post-contrast administration
Measure: Number; unit: Standard Uptake Value Ratio (SUVR)
Groups:
- Subject 201-0001; Subject 201-0002; Subject 201-0003; Subject 201-0004; Subject 201-0005; Subject 201-0006; Subject 201-0007: [18F]flutemetamol Injection-less than 10µg of flutemetamol.
Arm/Group | Subject 201-0001 | Subject 201-0002 | Subject 201-0003 | Subject 201-0004 | Subject 201-0005 | Subject 201-0006 | Subject 201-0007
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1
Standard Uptake Value Ratio (SUVR)
  Brain Region-Cerebellum-VOI surrounding biopsy | 1.59 | 1.56 | 1.25 | 2.17 | 2.07 | 1.39 | 1.00
  Brain Region-Cerebellum-Contralateral biopsy | 1.77 | 1.93 | 1.16 | 2.32 | 2.08 | 1.18 | 0.86
  Brain Region-Cerebellum-Anterior Cingulate | 2.19 | 2.36 | 1.44 | 2.81 | 2.65 | 1.26 | 1.27
  Brain Region-Cerebellum-Frontal Cortex | 2.24 | 2.78 | 1.32 | 2.71 | 2.74 | 1.28 | 1.19
  Brain Region-Cerebellum-Lateral Temporal Cortex | 2.08 | 2.35 | 1.45 | 2.56 | 2.63 | 1.52 | 1.32
  Brain Region-Cerebellum-Parietal Cortex | 1.99 | 2.38 | 1.38 | 2.84 | 2.27 | 1.36 | 1.35
  Brain Region-Cerebellum-Posterior Cortex | 2.11 | 2.33 | 1.40 | 2.86 | 2.73 | 1.17 | 1.73
  Brain Region-Cerebellum-Composite VOI | 2.13 | 2.48 | 1.39 | 2.74 | 2.62 | 1.34 | 1.34

2. Primary Outcome: Comparsion Between Brain Uptake of [18F] Flutemetamol Amyloid Level From Immunohistochemistry Assay and a Stained Biopsy Tissue Specimen.
Description: This was an amyloid level estimate measured by Immunohistochemistry assay to determine the percentage of plaque area for mAb NAB228. The Immuno-histo chemical reagent was monoclonal antibody (mAB) NAB228. This is a percentage of the area of the biopsy tissue specimen that stains positive for amyloid using NAB228.
Time Frame: Post-contrast administration
Measure: Number; unit: Percent plaque area
Groups:
- Subject 201-0001; Subject 201-0002; Subject 201-0003; Subject 201-0004; Subject 201-0005; Subject 201-0006; Subject 201-0007: [18F]flutemetamol Injection-(less than 10µg of flutemetamol).
Arm/Group | Subject 201-0001 | Subject 201-0002 | Subject 201-0003 | Subject 201-0004 | Subject 201-0005 | Subject 201-0006 | Subject 201-0007
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1
Percent plaque area | 0.127 | 0.447 | 0 | 1.007 | 0.4 | 0 | 0

3. Secondary Outcome: Quantitative Estimates of Amyloid Levels ( Percent % Plaque Load) for the Following 7 Subjects
Description: Using the Precent area of Plaque values from the Primary Anaylsis, determine the association between cerebral cortical uptake of [18F] flutemetamol (as contralateral, ipsilateral, and composite SUVR values) and Immunohistochemical and histochemical-based estimates of amyloid.
Time Frame: Post-contrast Administration
Population: Using the Precent area of Plaque values from the Primary Anaylsis, determine the association between cerebral cortical uptake of [18F] flutemetamol (as contralateral, ipsilateral, and composite SUVR values) and Immunohistochemical and histochemical-based estimates of amyloid.
Measure: Number; unit: Percentage of Plaque
Groups:
- Amyloid Level (Plaque Load): Amlyoid level estimate from the Immunohistochemistry assay: Percent plaque area (average across slides) for mAb NAB228.
Arm/Group | Amyloid Level (Plaque Load)
Number analyzed (Participants) | 7
Percentage of Plaque
  Subject-201-0001 | 0.127
  Subject-201-0002 | 0.447
  Subject-201-0003 | 0
  Subject-201-0004 | 1.007
  Subject-201-0005 | 0.4
  Subject-201-0006 | 0
  Subject-201-0007 | 0
Statistical Analysis 1: Comparison: Amyloid Level (Plaque Load); Contralateral to the biopsy Site; Test type: Non-Inferiority or Equivalence — The level of association between SUVR and the amyloid levels was analyzed using a regression model; p = 0.098, Regression, Linear; R² = 0.688
Statistical Analysis 2: Comparison: Amyloid Level (Plaque Load); Ipsilateral to the biopsy Site; Test type: Non-Inferiority or Equivalence — The level of association between SUVR and the amyloid levels was analyzed using a regression model; p = 0.268, Regression, Linear; R² = 0.482
Statistical Analysis 3: Comparison: Amyloid Level (Plaque Load); Composite Region; Test type: Non-Inferiority or Equivalence — The level of association between SUVR and the amyloid levels was analyzed using a regression model; p = 0.099, Regression, Linear; R² = 0.685

ADVERSE EVENTS:
Arm/Group | Flutemetamol Injection
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flutemetamol Injection (N=7)
Blood Pressure Increase (Investigations) | 5 (5)
Blood Glucose Decrease (Investigations) | 1 (1)
Dizziness (Investigations) | 1 (1)
Flushing (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No